CLINICAL TRIAL: NCT05402345
Title: A Phase II Randomized, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating Effect Of GlcNAc On Tear Production In Individuals With NGLY1-CDDG
Brief Title: A Study of GlcNAc on Tear Production in NGLY1-CDDG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eva Morava-Kozicz (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Eva Morava-Kozicz, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHOP 23-020868; 8404 (Other: FCDGC)
Record Dates: First submitted 2022-05-28; First posted 2022-06-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: NGLY1 Deficiency
MeSH Terms: conditions — NGLY1 deficiency | interventions — 4-O-(N-acetylglucosaminyl)glucosamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GlcNAc (Experimental): GlcNAc powder
  Interventions: Drug: GlcNAc-GlcN
- Placebo (Placebo Comparator): Placebo xylose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GlcNAc-GlcN — GlcNAc powder - weight-dependent dose
  Arms: GlcNAc
Other: Placebo — Placebo xylose
  Arms: Placebo

SUMMARY:
In patients with NGLY1-CDDG, the disorder can lead to eye damage due to not being able to produce enough tears. This study is being done to see if the dietary supplement, GlcNAc, improves tear production in patients with NGLY1-CDDG.

DETAILED DESCRIPTION:
This study is a multicenter randomized, double-blind, placebo-controlled trial of GlcNAc supplementation for improvement of tear production in NGLY1-CDDG. Clinical history and screening data will be reviewed to determine subject eligibility. If a subject is already on GlcNAc, a washout period of 1 month will be required prior to consent and randomization. Interested subjects who have a molecularly confirmed diagnosis of NGLY1-CDDG will be consented. Baseline data will be collected prior to randomization at treatment initiation. Subjects will then be randomized to placebo or GlcNAc. They will be administered weight-dependent doses of GlcNAc or an equivalent volume of placebo enterally for 6 weeks, followed by open label weight-dependent doses of GlcNAc for 6 weeks. A visit for evaluation and collection of lab samples will be conducted at 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Previously molecularly confirmed NGLY1-CDDG
* Between the ages of 1 year old to 60 years old
* Parent or legal guardian available to provide consent on behalf of minor subjects or adult subjects who are unable to give informed consent due to developmental disabilities. Willingness of subject or legal guardian to provide consent.
* Non-pregnant, non-lactating female subjects of childbearing potential who are heterosexually active must agree to use a highly effective method of contraception for the duration of the study. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly, such as oral/injectable/inserted/implanted/transdermal contraceptives, condom with diaphragm, condom with spermicide, diaphragm with spermicide, intrauterine hormone- releasing system, or intrauterine device (IUD), or sexual abstinence. Contraception is not required where at least 6 weeks have passed since sterilization, defined as females having undergone one of the following surgeries: hysterectomy, bilateral tubal ligation or occlusion, bilateral oophorectomy, or bilateral salpingectomy; and males who are vasectomized. Contraception is not required where females are postmenopausal (defined as 12 consecutive months of spontaneous amenorrhea and age ≥51 years)..

Exclusion Criteria

* Hypersensitivity to any of the components of the placebo
* History of treatment with GlcNAc within 28 days of Visit 1
* Participation in another therapeutic trial - the subject will not be permitted to participate in any other drug trial during the blinded phase and during the 28 days prior to Visit 1
* Shellfish allergy
* Planned eye surgery within 3 months of enrollment
* • Females that are pregnant, nursing or less than 6 months postpartum or attempting to conceive

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in tear production from baseline in placebo vs GlcNAc group | 6 weeks
  The primary endpoint of the study is the difference in tear production from baseline in individuals with NGLY1-CDDG between the placebo and the GlcNAc group after 6 weeks of blinded therapy, as measured by Schirmer II test which is a tool that helps assess the amount of tears in the eyes.

SECONDARY OUTCOMES:
Frequency of eye infections needing treatments | 6 weeks, 12 weeks
  Patient/family reported number of eye infections needing treatment in last month after 6 weeks of blinded therapy and at 12 weeks after 6 weeks of open-label administration of GlcNAc.
Frequency of eye redness needing treatments | 6 weeks, 12 weeks
  Patient/family reported frequency of eye redness after 6 weeks of blinded therapy and at 12 weeks after 6 weeks of open-label administration of GlcNAc.
Frequency of eye tearing/watering | 6 weeks, 12 weeks
  Patient/family reported frequency of eye tearing/watering after 6 weeks of blinded therapy and at 12 weeks after 6 weeks of open-label administration of GlcNAc.
Frequency of light sensitivity | 6 weeks, 12 weeks
  Patient/family reported frequency of light sensitivity after 6 weeks of blinded therapy and at 12 weeks after 6 weeks of open-label administration of GlcNAc.
Frequency of wind sensitivity | 6 weeks, 12 weeks
  Patient/family reported frequency of wind sensitivity after 6 weeks of blinded therapy and at 12 weeks after 6 weeks of open-label administration of GlcNAc.
Difference in tear production from baseline | 12 weeks
  Difference in tear production, as measured by Schirmer II test, at 12 weeks after 6 weeks of open-label administration of GlcNAc.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Morava-Kozicz, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No